CLINICAL TRIAL: NCT04671381
Title: Improving Access and Affordability of Adult Hearing Healthcare: Effectiveness of Community-based Interventions in West Central and South Alabama
Brief Title: Improving Access and Affordability of Adult Hearing Healthcare
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama, Tuscaloosa (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-03-2170
Record Dates: First submitted 2020-12-03; First posted 2020-12-17 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Correction of Hearing Impairment

STUDY DESIGN:
Intervention Model Description: Prior to the hearing evaluation, participants will be randomly placed in one of three groups. The three groups include those who will receive the current best practices care from an audiologist (ABP), those who will receive the ABP plus an aural rehabilitation program (ABP+AR), and finally, those who will receive only an OTC HA without assistance from an audiologist for providing programming, maintenance or care information (OTC-only). The AR programming will be provided by trained Community Health Advisors (CHAs). Both the ABP and OTC-only groups initially will attend general health information sessions in-place of the AR program. Once the ABP+AR groups have completed their AR sessions, the ABP and the OTC-only groups will attend the AR programming sessions. By using this service-delivery model, it will be possible to analyze the effectiveness of the AR programming, separate from any benefits that might occur simply by meeting with others in a group setting.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participant randomization will occur by generating three groups of random participant numbers and then assigning each participant to their designated group. Only the PI and the project manager will have access to the randomization lists. The PI will generate the randomization lists and the Project Manager will assign the participants accordingly to each group. Audiologists will be blinded to the intervention condition for participants. Specifically, two audiologists (A1 and A2) will conduct the initial hearing evaluations. A2 will perform the OTC HA settings and orientations and a third audiologist (A3) will perform the follow-up speech perception testing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Audiology Best Practices plus Aural Rehabilitation (ABP+AR) (Experimental): This experimental group will receive a hearing evaluation, an over-the-counter hearing aid fitting and orientation, and four-weeks of an aural rehabilitation program conducted by specially-trained community health workers. Additionally, these adults will complete pre- and post-questionnaires and speech perception testing.
  Interventions: Behavioral: Hearing Evaluation; Device: Over-the-Counter Hearing Aid (OTC HA) Fitting and Orientation; Behavioral: Four Weeks of Aural Rehabilitation
- Audiology Best Practices (ABP) (Active Comparator): This comparison group of adults with hearing loss will receive a hearing evaluation and over-the-counter hearing aid fitting and orientation. The aural rehabilitation program will not be provided initially. These participants will complete pre- and post-questionnaires and speech perception testing.
  Interventions: Behavioral: Hearing Evaluation; Behavioral: Four Weeks of Aural Rehabilitation
- Over-the-Counter Only (OTC-Only) (Active Comparator): This comparison group of adults with hearing loss will receive a hearing evaluation. They will be provided with over-the-counter hearing aids but the audiologist will not assist with fitting the aids or providing an orientation. This arm mimics what would happen when a consumer privately purchases over-the-counter hearing aids. They will complete pre- and post-questionnaires and speech perception testing.
  Interventions: Behavioral: Hearing Evaluation; Device: Provision of Over-the-Counter Hearing Aids

INTERVENTIONS:
Behavioral: Hearing Evaluation — Behavioral thresholds for pure tones will be conducted along with speech perception measures.
Device: Over-the-Counter Hearing Aid (OTC HA) Fitting and Orientation — Study participants will be fitted with binaural OTC HAs in addition to receiving information on how to use and care for their devices.
  Other Names: Over-the-Counter Hearing Aid Fitting and Orientation
  Arms: Audiology Best Practices plus Aural Rehabilitation (ABP+AR)
Behavioral: Four Weeks of Aural Rehabilitation — Participants will receive four weeks of information sessions to help them adjust to their over-the-counter hearing aid and their hearing loss.
  Arms: Audiology Best Practices (ABP); Audiology Best Practices plus Aural Rehabilitation (ABP+AR)
Device: Provision of Over-the-Counter Hearing Aids — Study participants will receive binaural OTC HAs. Participants will fit their OTC HAs based on manufacturer guidelines without the help of an audiologist.
  Other Names: Provision of Over-the Counter Hearing Aids
  Arms: Over-the-Counter Only (OTC-Only)

SUMMARY:
This project will address quality of care issues associated with hearing loss in adults who have mild-to-moderate hearing loss and who have no access to hearing healthcare. Through the use of three different interventions involving over-the-counter hearing aids, it will lead to options that will increase access and affordability of hearing healthcare for adults with mild-to-moderate hearing loss.

DETAILED DESCRIPTION:
The design for this study is outlined below according to each Aim.

Aim 1: To identify the effectiveness of over-the-counter hearing aids (OTC HAs) for decreasing hearing handicap and improving speech perception in adults with no access to hearing health care.

Aim 2: To implement an adult aural rehabilitation (AR) program for those without access to hearing health care to improve OTC HA benefit, promote OTC HA use and lead to increased quality of life (QOL).

Aim 1 will assess the effectiveness of OTC HAs for our participant population and Aim 2 will implement an AR program. With Aim 1, hearing loss will be assessed and an OTC HA will be provided. Prior to the hearing evaluation, participants will be randomly placed in one of three groups to assess the effectiveness of the AR program (Aim 2). The three groups include those who will receive the current best practices care from an audiologist (ABP), those who will receive the ABP plus an aural rehabilitation program (ABP+AR), and finally, those who will receive only an OTC HA without assistance from an audiologist for providing programming, maintenance or care information (OTC-only). Both the ABP and OTC-only groups initially will attend general health information sessions in-place of the AR program. Local health care providers who have training in general health areas such as nutrition, diabetes, obesity, and heart health to name a few, will provide the General Health and Wellness programming. Once the ABP+AR groups have completed their AR sessions, the ABP and the OTC-only groups will attend the AR programming sessions. This testing layout and schedule is provided in the table below.

Randomization will occur for each county visited and for the participants. Specifically, five counties will each receive a code and these codes will be randomized to determine when the study will take place in that area. All five regions will be included over a one-year period. Participant randomization will occur by generating three groups of random participant numbers and then assigning each participant to their designated group. Only the PI and the project manager will have access to the randomization lists. The PI will generate the randomization lists and the Project Manager will assign the participants accordingly to each group. The randomization lists will be kept on a password-protected computer and only accessible by the PI or Project Manager.

Audiologists will be blinded to the intervention condition for participants. Specifically, two audiologists (A1 and A2) will conduct the initial hearing evaluations. A2 will perform the OTC HA settings and orientations and a third audiologist (A3) will perform the follow-up speech perception testing in weeks 8 - 9. A second post-speech perception testing for all participants in week 14 will be conducted by A1.

The entire program will take place over a 14-week period for one county at a time. County 1 will begin at Week 1 and the remaining four regions will be stratified such that testing will begin at Week 9, 10 or 11 consecutively for each region. The stratification will be done to ensure that testing takes place in each area over a one-year period, and also, to avoid simultaneous testing at two sites. Finally, all participants who complete the study in years 1 and 2 will be invited back to complete speech perception testing and the AR surveys one year after they complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Mild-to-moderate hearing loss
* Live in West Central or South Alabama
* 40 years of age or older

Exclusion Criteria:

• Medical conditions resulting in severe cognitive impairment (e.g., stroke, head injury, senile dementia or Alzheimer's disease)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Measuring Change in the Hearing Handicap Inventory for Elderly (HHIE) Outcomes | A baseline outcome will be obtained prior to over-the-counter hearing aid fitting. Outcomes will be measured at weeks 4 to 7 of intervention, during week 14 of the intervention, and through study completion, or 1 assessment each year.
  Twenty-five questions of the Hearing Handicap Inventory for Elderly (HHIE) measure emotional and social/situational consequences of hearing loss, including feelings of embarrassment, social isolation, and frustration. Scores range from 0 to 100 with higher scores indicative of poorer performance.
Measuring Change in International Outcome Inventory for Hearing Aids (IOI-HA) Outcomes | A baseline outcome will be obtained prior to over-the-counter hearing aid fitting. Outcomes will be measured at weeks 4 to 7 of intervention, during week 14 of the intervention, and through study completion, or 1 assessment each year.
  The International Outcome Inventory for Hearing Aids (IOI-HA) is an eight-item inventory that assesses daily use of over-the-counter hearing aid use, over-the-counter hearing aid benefit, and activity limitations to name a few. This is a scaled qualitative measure that assesses outcomes over time.

SECONDARY OUTCOMES:
Measuring Change in Northwestern University-6 (NU-6) Word Recognition Outcomes | A baseline outcome will be obtained prior to over-the-counter hearing aid fitting. Outcomes will be measured at weeks 8 to 9 of intervention, during week 14 of the intervention, and through study completion, or 1 assessment each year.
  This test will assess word recognition in quiet. Binaural testing will be performed at 65 dBA in the sound field. A percentage correct word understanding will be obtained. A higher scores is indicative of better performance.
Measuring Change in Quick Speech In Noise (SIN) Word Recognition Outcomes | A baseline outcome will be obtained prior to over-the-counter hearing aid fitting. Outcomes will be measured at weeks 8 to 9 of intervention, during week 14 of the intervention, and through study completion, or 1 assessment each year.
  The participant will be instructed to repeat the presented sentences in noise via a speaker presented at 0˚ azimuth. The correctly identified target words will be totaled and then subtracted from 25.5 to obtain the Signal-to-Noise Ratio (SNR) loss. A higher score is indicative of poorer performance.
Measuring Change in the Client Oriented Scale of Improvement (COSI) | A baseline outcome will be obtained prior to over-the-counter hearing aid fitting. Outcomes will be measured at weeks 4 to 7 of intervention, during week 14 of the intervention, and through study completion, or 1 assessment each year.
  The Client Oriented Scale of Improvement (COSI) is a 16-item clinician-administered survey that addresses how the participants' five most important listening difficulties have been alleviated with over-the-counter hearing aid use. This is a qualitative scale that measures improvement over time.
Measuring Change in the Abbreviated Profile of Hearing Aid Benefit (APHAB) | A baseline outcome will be obtained prior to over-the-counter hearing aid fitting. Outcomes will be measured at weeks 4 to 7 of intervention, during week 14 of the intervention, and through study completion, or 1 assessment each year.
  The Abbreviated Profile of Hearing Aid Benefit (APHAB) is a 24-item survey that computes OTC HA-benefit by calculating the difference between aided and unaided conditions. It is a qualitative scale that measures the extent of change over time.
Measuring Change in the World Health Organization Quality of Life-Age (WHOQOL-AGE) Survey | A baseline outcome will be obtained prior to over-the-counter hearing aid fitting. Outcomes will be measured at weeks 4 to 7 of intervention, during week 14 of the intervention, and through study completion, or 1 assessment each year.
  The World Health Organization Quality of Life-Age (WHOQOL-AGE) survey is a 13-item scale that examines quality of life in adults as they age. It is a qualitative rating scale that can help to identify change in performance over time.

CONTACTS AND LOCATIONS:
Overall Officials: Marcia J Hay-McCutcheon, PhD, Principal Investigator — The University of Alabama, Tuscaloosa
Locations (1):
- The University of Alabama, Tuscaloosa, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data that has been collected during this clinical trial and after it has been de-identified will be shared.
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 3 months following article publication and ending 5 years after the article has been published.
Access Criteria: Researchers who provide a methodologically sound proposal will be given access to the data.

REFERENCES:
- [Result] Tillman TW, Carhart R. An expanded test for speech discrimination utilizing CNC monosyllabic words. Northwestern University Auditory Test No. 6. SAM-TR-66-55. Tech Rep SAM-TR. 1966 Jun:1-12. doi: 10.21236/ad0639638. No abstract available. PMID 5296571
- [Result] Schow RL, Nerbonne MA. Communication screening profile: use with elderly clients. Ear Hear. 1982 May-Jun;3(3):135-47. doi: 10.1097/00003446-198205000-00007. No abstract available. PMID 7095322
- [Result] Cox RM, Alexander GC. The International Outcome Inventory for Hearing Aids (IOI-HA): psychometric properties of the English version. Int J Audiol. 2002 Jan;41(1):30-5. doi: 10.3109/14992020209101309. PMID 12467367
- [Result] Dillon H, James A, Ginis J. Client Oriented Scale of Improvement (COSI) and its relationship to several other measures of benefit and satisfaction provided by hearing aids. J Am Acad Audiol. 1997 Feb;8(1):27-43. PMID 9046067
- [Result] Cox RM, Alexander GC. The abbreviated profile of hearing aid benefit. Ear Hear. 1995 Apr;16(2):176-86. doi: 10.1097/00003446-199504000-00005. PMID 7789669
- [Result] Caballero FF, Miret M, Power M, Chatterji S, Tobiasz-Adamczyk B, Koskinen S, Leonardi M, Olaya B, Haro JM, Ayuso-Mateos JL. Validation of an instrument to evaluate quality of life in the aging population: WHOQOL-AGE. Health Qual Life Outcomes. 2013 Oct 23;11:177. doi: 10.1186/1477-7525-11-177. PMID 24152691
- [Result] Etymotic. QuickSIN Speech-in-Noise Test. Elk Grove Village, IL 2006.
- [Derived] Hay-McCutcheon MJ, Hubbard A, Brothers EB, Straub K, Allen RS, Hardy C, Tye-Murray N. Development and Implementation of an Aural Rehabilitation Program Using Community Health Workers in Rural Alabama. Perspect ASHA Spec Interest Groups. 2024 Oct;9(5):1367-1376. doi: 10.1044/2024_PERSP-24-00083. Epub 2024 Aug 28. PMID 40123580

DOCUMENTS (1):
  • Informed Consent Form (2024-07-26): https://cdn.clinicaltrials.gov/large-docs/81/NCT04671381/ICF_004.pdf